CLINICAL TRIAL: NCT00753545
Title: Phase II Randomised, Double Blind, Multicentre Study to Assess the Efficacy of AZD2281 in the Treatment of Patients With Platinum Sensitive Relapsed Serous Ovarian Cancer Following Treatment With Two or More Platinum Containing Regimens
Brief Title: Assessment of Efficacy of AZD2281 in Platinum Sensitive Relapsed Serous Ovarian Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D0810C00019; 2008-003439-18 (EudraCT Number)
Expanded Access: NCT03079687 (Approved for marketing)
Record Dates: First submitted 2008-09-12; First posted 2008-09-16 (Estimated); Results first posted 2013-03-11 (Estimated); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Ovarian Cancer
Keywords: Serous,; Ovarian cancer,; PARP,; BRCA1,; BRCA2,; Poly(ADP ribose) polymerases,; Platinum sensitive,; Homologous Recombination Deficiency (HRD)
MeSH Terms: conditions — Ovarian Neoplasms; Fanconi Anemia, Complementation Group D1 | interventions — olaparib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): AZD2281
  Interventions: Drug: AZD2281
- 2 (Placebo Comparator): matching placebo
  Interventions: Drug: matching placebo

INTERVENTIONS:
Drug: AZD2281 — Tablets Oral BID
  Other Names: Olaparib, Lynparza
  Arms: 1
Drug: matching placebo — matching placebo bid
  Arms: 2

SUMMARY:
The primary purpose of this study to determine if AZD2281 is effective and well tolerated in maintaining the improvement in your cancer after previous platinum-based chemotherapy

ELIGIBILITY:
Inclusion Criteria:

* Female patients with histologically diagnosed serous ovarian cancer or recurrent serous ovarian cancer.
* Patients must have completed at least 2 previous courses of platinum containing therapy; the patient must have been platinum sensitive to the penultimate chemo regimen.
* For the last chemotherapy course prior to enrolment on the study, patients must have demonstrated an objective stable maintained response (partial or complete response) and this response needs to be maintained until completion of chemotherapy.
* Patients must be treated on the study within 8 wks of completion of their final dose of the platinum containing regimen.

Exclusion Criteria:

* Previous treatment with PARP inhibitors including AZD2281
* Patients with low grade ovarian carcinoma.
* Patients who have had drainage of their ascites during the final 2 cycles of their last chemotherapy regimen prior to enrolment on the study
* Patients receiving any chemotherapy, radiotherapy (except for palliative reasons), within 2 weeks from the last dose prior to study entry (or a longer period depending on the defined characteristics of the agents used).

Ages: 18 Years to 130 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 265 (Actual)
Dates: Start 2008-08-28 (Actual); Primary Completion 2010-06-30 (Actual); Study Completion 2023-10-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mika Sovak, BSc, MBCHB, MD, Study Director — AstraZeneca; Prof Jonathan A Lederman, Principal Investigator — University College, London
Locations (92):
- United States (9):
  - Research Site, Berkeley, California
  - Research Site, San Francisco, California
  - Research Site, West Hollywood, California
  - Research Site, Sunrise, Florida
  - Research Site, West Palm Beach, Florida
  - Research Site, Indianapolis, Indiana
  - Research Site, Boston, Massachusetts
  - Research Site, New York, New York
  - Research Site, Providence, Rhode Island
- Australia (8):
  - Research Site, Adelaide
  - Research Site, East Bentleigh
  - Research Site, Heidelberg
  - Research Site, Melbourne
  - Research Site, Nambour
  - Research Site, Randwick
  - Research Site, South Brisbane
  - Research Site, Toorak Gardens
- Austria (3):
  - Research Site, Innsbruck
  - Research Site, Vienna
  - Research Site, Wein
- Belgium (2):
  - Research Site, Brussels
  - Research Site, Leuven
- Canada (4):
  - Research Site, Vancouver, British Columbia
  - Research Site, Toronto, Ontario
  - Research Site, Québec, Quebec
  - Research Site, Sherbrooke, Quebec
- Czechia (3):
  - Research Site, Brno
  - Research Site, Olomouc
  - Research Site, Prague
- Estonia (2):
  - Research Site, Tallinn
  - Research Site, Tartu
- France (6):
  - Research Site, Bordeaux
  - Research Site, Caen
  - Research Site, Lyon
  - Research Site, Nantes
  - Research Site, Paris
  - Research Site, Reims
- Germany (12):
  - Research Site, Bonn
  - Research Site, Düsseldorf
  - Research Site, Essen
  - Research Site, Freiburg im Breisgau
  - Research Site, Göttingen
  - Research Site, Hanover
  - Research Site, Kiel
  - Research Site, Marburg
  - Research Site, München
  - Research Site, Rostock
  - Research Site, Ulm
  - Research Site, Wiesbaden
- Israel (7):
  - Research Site, Haifa
  - Research Site, Holon
  - Research Site, Jerusalem
  - Research Site, Nahariya
  - Research Site, Ramat Gan
  - Research Site, Tel Aviv
  - Research Site, Ẕerifin
- Research Site, Amsterdam, Netherlands
- Poland (6):
  - Research Site, Bialystok
  - Research Site, Grzepnica
  - Research Site, Lublin
  - Research Site, Poznan
  - Research Site, Szczecin
  - Research Site, Warsaw
- Romania (4):
  - Research Site, Baia Mare
  - Research Site, Cluj-Napoca
  - Research Site, Iași
  - Research Site, Suceava
- Russia (8):
  - Research Site, Barnaul
  - Research Site, Obninsk
  - Research Site, Orenburg
  - Research Site, Perm
  - Research Site, Pyatigorsk
  - Research Site, Saint Petersburg
  - Research Site, Voronezh
  - Research Site, Yekaterinburg
- Spain (3):
  - Research Site, Córdoba
  - Research Site, Madrid
  - Research Site, Valencia
- Ukraine (7):
  - Research Site, Donetsk
  - Research Site, Kharkiv Region
  - Research Site, Kyiv
  - Research Site, Lutsk
  - Research Site, Odesa
  - Research Site, Ternopil
  - Research Site, Uzhhorod
- United Kingdom (7):
  - Research Site, Dundee
  - Research Site, Edinburgh
  - Research Site, London
  - Research Site, Manchester
  - Research Site, Metropolitan Borough of Wirral
  - Research Site, Northwood
  - Research Site, Sutton

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Barnicle A, Ray-Coquard I, Rouleau E, Cadoo K, Simpkins F, Aghajanian C, Leary A, Poveda A, Lheureux S, Pujade-Lauraine E, You B, Ledermann J, Matulonis U, Gourley C, Timms KM, Lai Z, Hodgson DR, Elks CE, Dearden S, Egile C, Lao-Sirieix P, Harrington EA, Brown JS. Patterns of genomic instability in > 2000 patients with ovarian cancer across six clinical trials evaluating olaparib. Genome Med. 2024 Dec 18;16(1):145. doi: 10.1186/s13073-024-01413-5. PMID 39695768
- [Derived] Tattersall A, Ryan N, Wiggans AJ, Rogozinska E, Morrison J. Poly(ADP-ribose) polymerase (PARP) inhibitors for the treatment of ovarian cancer. Cochrane Database Syst Rev. 2022 Feb 16;2(2):CD007929. doi: 10.1002/14651858.CD007929.pub4. PMID 35170751
- [Derived] Ledermann JA, Harter P, Gourley C, Friedlander M, Vergote I, Rustin G, Scott C, Meier W, Shapira-Frommer R, Safra T, Matei D, Fielding A, Bennett B, Parry D, Spencer S, Mann H, Matulonis U. Quality of life during olaparib maintenance therapy in platinum-sensitive relapsed serous ovarian cancer. Br J Cancer. 2016 Nov 22;115(11):1313-1320. doi: 10.1038/bjc.2016.348. Epub 2016 Nov 8. PMID 27824811
- [Derived] Ledermann JA, Harter P, Gourley C, Friedlander M, Vergote I, Rustin G, Scott C, Meier W, Shapira-Frommer R, Safra T, Matei D, Fielding A, Spencer S, Rowe P, Lowe E, Hodgson D, Sovak MA, Matulonis U. Overall survival in patients with platinum-sensitive recurrent serous ovarian cancer receiving olaparib maintenance monotherapy: an updated analysis from a randomised, placebo-controlled, double-blind, phase 2 trial. Lancet Oncol. 2016 Nov;17(11):1579-1589. doi: 10.1016/S1470-2045(16)30376-X. Epub 2016 Sep 9. PMID 27617661
- [Derived] Matulonis UA, Harter P, Gourley C, Friedlander M, Vergote I, Rustin G, Scott C, Meier W, Shapira-Frommer R, Safra T, Matei D, Fielding A, Spencer S, Parry D, Grinsted L, Ledermann JA. Olaparib maintenance therapy in patients with platinum-sensitive, relapsed serous ovarian cancer and a BRCA mutation: Overall survival adjusted for postprogression poly(adenosine diphosphate ribose) polymerase inhibitor therapy. Cancer. 2016 Jun 15;122(12):1844-52. doi: 10.1002/cncr.29995. Epub 2016 Apr 8. PMID 27062051
- [Derived] Ledermann J, Harter P, Gourley C, Friedlander M, Vergote I, Rustin G, Scott CL, Meier W, Shapira-Frommer R, Safra T, Matei D, Fielding A, Spencer S, Dougherty B, Orr M, Hodgson D, Barrett JC, Matulonis U. Olaparib maintenance therapy in patients with platinum-sensitive relapsed serous ovarian cancer: a preplanned retrospective analysis of outcomes by BRCA status in a randomised phase 2 trial. Lancet Oncol. 2014 Jul;15(8):852-61. doi: 10.1016/S1470-2045(14)70228-1. Epub 2014 May 31. PMID 24882434
- [Derived] Ledermann J, Harter P, Gourley C, Friedlander M, Vergote I, Rustin G, Scott C, Meier W, Shapira-Frommer R, Safra T, Matei D, Macpherson E, Watkins C, Carmichael J, Matulonis U. Olaparib maintenance therapy in platinum-sensitive relapsed ovarian cancer. N Engl J Med. 2012 Apr 12;366(15):1382-92. doi: 10.1056/NEJMoa1105535. Epub 2012 Mar 27. PMID 22452356
- [Derived] Yap TA, Carden CP, Kaye SB. Beyond chemotherapy: targeted therapies in ovarian cancer. Nat Rev Cancer. 2009 Mar;9(3):167-81. doi: 10.1038/nrc2583. PMID 19238149
- See also: CSR_Synopsis_Redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D0810C00019&attachmentIdentifier=e1c8bfef-5d82-4db6-adaa-bd261623eaf8&fileName=CSR_Synopsis_Redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first patient was enrolled on 28 August 2008 and the last patient was enrolled on 9 February 2010. Patients were enrolled at 82 centres in 16 countries. Of the 326 patients enrolled, 265 were randomized
Pre-assignment Details: It was planned that 250 women with advanced platinum sensitive serous ovarian cancer who had received 2 or more previous platinum-containing regimens and demonstrated an objective stable maintained response in the last platinum regimen prior to enrolment were to receive olaparib 400 mg bd or matching placebo in a 1:1 ratio. 265 randomised.
Groups:
- Olaparib 400 mg bd: AZD2281 olaparib (AZD2281) 400 mg oral capsules twice daily
- Placebo bd: olaparib matching placebo oral capsules twice daily
Period: Overall Study
Arm/Group | Olaparib 400 mg bd | Placebo bd
Started | 136 (Patients randomized) | 129 (Patients randomized)
Completed | 28 (Patients completing the Study) | 11 (Patients completing the Study)
Not Completed | 108 | 118
Not completed — Death | 98 | 112
Not completed — Lost to Follow-up | 2 | 3
Not completed — Protocol Violation | 1 | 0
Not completed — Voluntary Discontinuation of Patient | 7 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Olaparib 400 mg bd | Placebo bd | Total
Number analyzed (Participants) | 136 | 129 | 265
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.9 (10.95) | 58.5 (9.89) | 58.7 (10.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 136 | 129 | 265
  Male | 0 | 0 | 0
Time to progression [Number; unit: participants] — The time to disease progression from the completion of the penultimate platinum containing therapy (last dose) prior to enrolment on the study.
  participants
    >6 to 12 months | 53 | 54 | 107
    >12 months | 83 | 75 | 158
Objective response [Number; unit: Participants] — Objective response to the last platinum containing regimen prior to enrolment on the study:
  * CR-Complete Response (defined as normal radiological findings and CA-125 within the normal range)
  * PR-Partial Response (defined as a RECIST PR and/or GCIG CA-125 response)
  Participants
    Complete response | 57 | 63 | 120
    Partial response | 79 | 66 | 145

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS) (According to Response Evaluation Criteria in Solid Tumours [RECIST])
Description: PFS was defined as the time from randomisation to the earlier date of radiological progression (per RECIST criteria) or death by any cause in the absence of objective progression. [Full analysis set (FAS)]
Time Frame: Radiologic scans performed at baseline then every 12 weeks (+/- 1 week) for the first 60 weeks, then every 24 weeks (+/-1 week) thereafter, assessed maximum up to 14 months.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Olaparib 400 mg bd | Placebo bd
Number analyzed (Participants) | 136 | 129
Months | 8.4 [7.4 to 11.5] | 4.8 [4.0 to 5.5]
Statistical Analysis 1: Comparison: Olaparib 400 mg bd vs Placebo bd; HR < 1 favours olaparib; Test type: Superiority or Other; p < 0.00001, Regression, Cox; The model includes factors for treatment, ethnic descent, platinum sensitivity and response to final platinum therapy; Hazard Ratio (HR) = 0.35, 95% CI 2-sided [0.25 to 0.49]

2. Secondary Outcome: Overall Survival (OS)
Description: OS = time from randomisation to date of death from any cause. Patients who had not died at time of analysis were censored at last date patient was known to be alive.
Time Frame: Follow up every 12 weeks post progression, assessed maximum up to 90 months.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Olaparib 400 mg bd | Placebo bd
Number analyzed (Participants) | 136 | 129
Months | 29.8 [26.9 to 35.7] | 27.8 [24.9 to 33.7]
Statistical Analysis 1: Comparison: Olaparib 400 mg bd vs Placebo bd; HR < 1 favours olaparib; Test type: Superiority or Other; p = 0.02, Regression, Cox; The model includes factors for treatment, ethnic descent, platinum sensitivity and response to final platinum therapy; Hazard Ratio (HR) = 0.73, 95% CI 2-sided [0.55 to 0.95]

3. Secondary Outcome: Objective Response Rate (ORR) (According to RECIST)
Description: For each treatment group, the ORR was the number of Complete Response (CR) and Partial Response (PR) divided by the number of patients in the group in the FAS with measurable disease at baseline (displayed as a percentage below). Evaluable for response set
Time Frame: as for outcome 1
Population: Evaluable for response set - A subset of the full analysis set which includes patients with measurable disease at baseline
Measure: Number; unit: percentage of participants
Arm/Group | Olaparib 400 mg bd | Placebo bd
Number analyzed (Participants) | 57 | 48
percentage of participants | 12.3 | 4.2

4. Secondary Outcome: Disease Control Rate
Description: Disease control rate was defined as the percentage of patients who have at least 1 confirmed visit response of CR or PR or have demonstrated SD or NED for at least 23 weeks (ie, 24 weeks +/- 1 week) prior to any evidence of progression. [FAS]
Time Frame: Assessed at 24 weeks. Radiologic scans performed at baseline, week 12 (+/- 1 week) and week 24 (+/- 1 week).
Measure: Number; unit: percentage of participants
Arm/Group | Olaparib 400 mg bd | Placebo bd
Number analyzed (Participants) | 136 | 129
percentage of participants | 53.7 | 25.6

5. Secondary Outcome: Duration of Response
Description: Duration of response = time from assessment prior to timepoint where PR or CR confirmed (i.e. initial assessment of PR/CR), until earliest date of objective progression or death. [Responding patients only]. There were insufficient responses to enable conclusions to be drawn.
Time Frame: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Olaparib 400 mg bd | Placebo bd
Number analyzed (Participants) | 136 | 129
Months | 4.2 [2.8 to 5.6] | 2.3 [1.8 to 2.8]

6. Secondary Outcome: Percentage Change From Baseline in Tumour Size at Week 24
Description: Percentage change from baseline to Week 24 in target tumour size.
Time Frame: Radiologic scans performed at baseline then every 12 weeks (+/- 1week) for the first 60 weeks, then every 24 weeks (+/-1 week) thereafter, assessed maximum up to 14 months.
Population: as for outcome 3
Measure: Least Squares Mean (Full Range); unit: Percent change in tumour size
Arm/Group | Olaparib 400 mg bd | Placebo bd
Number analyzed (Participants) | 56 | 47
Percent change in tumour size | -0.8 [-100.0 to 45.0] | 26.4 [-36.4 to 39.4]
Statistical Analysis 1: Comparison: Olaparib 400 mg bd vs Placebo bd; LS mean < 0 favours olaparib; Test type: Superiority or Other; p = 0.03185, ANCOVA; The model includes factors for treatment, ethnic descent, platinum sensitivity and response to final platinum therapy; Difference in LS means = -27.1, 95% CI 2-sided [-51.9 to -2.4]

7. Secondary Outcome: Best Percentage Change in Cancer Antigen 125 (CA-125) Levels
Description: Best percentage change from baseline in CA-125 level
Time Frame: CA-125 was measured at baseline then every 28 days on treatment, assessed maximum up to 14 months.
Population: A subset of the FAS with baseline and at least 1 follow-up value of CA-125
Measure: Median (Full Range); unit: percentage of change
Arm/Group | Olaparib 400 mg bd | Placebo bd
Number analyzed (Participants) | 135 | 128
percentage of change | -16.67 [-100.00 to 346.15] | 0.00 [-99.50 to 1436.84]

8. Secondary Outcome: Best Objective Response
Description: Best overall response from radiologic assessments. [FAS]
Time Frame: Radiologic scans performed at baseline then every 12 weeks (+/- 1week) for the first 60 weeks, then every 24 weeks (+/- 1 week) thereafter, assessed maximum up to 14 months.
Measure: Number; unit: Participants
Arm/Group | Olaparib 400 mg bd | Placebo bd
Number analyzed (Participants) | 136 | 129
Participants
  Complete Response | 0 | 0
  Partial Response | 7 | 2
  No evidence of disease | 49 | 42
  Stable Disease >= 11 weeks | 46 | 25
  Disease Progression | 24 | 55
  Not Evaluable | 10 | 5

9. Secondary Outcome: RECIST and CA-125 Response Separately and Combined
Description: RECIST and CA-125 response separately and combined [Patients evaluable for either CA-125 response or RECIST response]
Time Frame: Radiologic scans performed at baseline then every 12 weeks (+/- 1week) for the first 60 weeks, then every 24 weeks (+/- 1 week) thereafter and monthly for CA-125 measurements, assessed maximum up to 14 months.
Measure: Number; unit: Participants
Arm/Group | Olaparib 400 mg bd | Placebo bd
Number analyzed (Participants) | 61 | 53
Participants
  RECIST Response | 16 | 2
  Confirmed RECIST Response | 7 | 2
  Unconfirmed RECIST response | 9 | 0
  CA-125 Response | 1 | 1
  Confirmed RECIST or CA-125 Response | 8 | 3

10. Secondary Outcome: Time to Earlier of CA-125 or RECIST Progression
Description: Time from randomisation to the earlier date of radiological progression (per RECIST criteria) or CA-125 or death by any cause in the absence of objective progression. [FAS]
Time Frame: Radiologic scans performed at baseline then every 12 weeks (+/- 1 week) for the first 60 weeks, then every 24 weeks (+/- 1 week) thereafter and monthly for CA-125 measurements, assessed maximum up to 14 months.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Olaparib 400 mg bd | Placebo bd
Number analyzed (Participants) | 136 | 129
Months | 8.3 [5.5 to 10.3] | 3.7 [2.8 to 4.5]
Statistical Analysis 1: Comparison: Olaparib 400 mg bd vs Placebo bd; HR < 1 favours olaparib; Test type: Superiority or Other; p < 0.00001, Regression, Cox; The model includes factors for treatment, ethnic descent, platinum sensitivity and response to final platinum therapy; Hazard Ratio (HR) = 0.35, 95% CI 2-sided [0.25 to 0.47]

11. Secondary Outcome: Improvement Rate for FACT-O Symptom Index (FOSI)
Description: The percentage of patients with an improvement in FOSI. Improvement was defined as a change from baseline of greater than or equal to +3. [Evaluable for FOSI set]
Time Frame: Patient reported outcome questionnaire completed at baseline then every 28 days up to disease progression, assessed maximum up to 14 months.
Population: Evaluable for FOSI set - A subset of the full analysis set which includes patients who have evaluable QoL/Symptom Endpoints at baseline
Measure: Number; unit: percentage of evaluable participants
Arm/Group | Olaparib 400 mg bd | Placebo bd
Number analyzed (Participants) | 117 | 115
percentage of evaluable participants | 17.1 | 14.8

12. Secondary Outcome: Improvement Rate for Trial Outcome Index (TOI)
Description: The percentage of patients with an improvement in TOI. Improvement was defined as a change from baseline of greater than or equal to +7. [Evaluable for TOI set]
Time Frame: as for outcome 11
Population: Evaluable for TOI - a subset of the full analysis set which includes patients who have evaluable QoL/Symptom Endpoints at baseline
Measure: Number; unit: percentage of evaluable participants
Arm/Group | Olaparib 400 mg bd | Placebo bd
Number analyzed (Participants) | 115 | 111
percentage of evaluable participants | 20.0 | 18.0

13. Secondary Outcome: Improvement Rate for Total Functional Analysis of Cancer Therapy - Ovarian (FACT-O)
Description: The percentage of patients with an improvement in total FACT-O. Improvement was defined as a change from baseline of greater than or equal to +9. [Evaluable for FACT-O set]
Time Frame: as for outcome 11
Population: Evaluable for Total Fact-O set - A subset of the full analysis set which includes patients who have evaluable QoL/Symptom Endpoints at baseline
Measure: Number; unit: percentage of evaluable participants
Arm/Group | Olaparib 400 mg bd | Placebo bd
Number analyzed (Participants) | 114 | 111
percentage of evaluable participants | 21.1 | 18.9

14. Secondary Outcome: FACT-O Symptom Index (FOSI) Time to Worsening
Description: The time to worsening was compared between treatments for each of the TOI, FOSI and total FACT-O. [Evaluable for FOSI set]
Time Frame: as for outcome 11
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Olaparib 400 mg bd | Placebo bd
Number analyzed (Participants) | 117 | 115
Months | 2.8 [1.8 to 3.7] | 3.7 [3.3 to 5.6]
Statistical Analysis 1: Comparison: Olaparib 400 mg bd vs Placebo bd; HR < 1 favours olaparib; Test type: Superiority or Other; p = 0.22, Regression, Cox; The model includes factors for treatment, ethnic descent, platinum sensitivity and response to final platinum therapy; Hazard Ratio (HR) = 1.23, 95% CI 2-sided [0.88 to 1.71]

15. Secondary Outcome: Trial Outcome Index(TOI)Time to Worsening
Description: The time to worsening was compared between treatments for each of the TOI, FOSI and total FACT-O. [Evaluable for TOI set]
Time Frame: as for outcome 11
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Olaparib 400 mg bd | Placebo bd
Number analyzed (Participants) | 115 | 111
Months | 3.8 [2.8 to 7.4] | 4.6 [3.7 to 7.4]
Statistical Analysis 1: Comparison: Olaparib 400 mg bd vs Placebo bd; HR < 1 favours olaparib; Test type: Superiority or Other; p = 0.67, Regression, Cox; The model includes factors for treatment, ethnic descent, platinum sensitivity and response to final platinum therapy; Hazard Ratio (HR) = 1.08, 95% CI 2-sided [0.75 to 1.56]

16. Secondary Outcome: Functional Analysis of Cancer Therapy - Ovarian (FACT-O) Time to Worsening
Description: The time to worsening was compared between treatments for each of the TOI, FOSI and total FACT-O. [Evaluable for FACT-O set]
Time Frame: as for outcome 11
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Olaparib 400 mg bd | Placebo bd
Number analyzed (Participants) | 114 | 111
Months | 2.8 [1.9 to 4.7] | 4.6 [3.6 to 5.5]
Statistical Analysis 1: Comparison: Olaparib 400 mg bd vs Placebo bd; HR < 1 favours olaparib; Test type: Superiority or Other; p = 0.38, Regression, Cox; The model includes factors for treatment, ethnic descent, platinum sensitivity and response to final platinum therapy; Hazard Ratio (HR) = 1.16, 95% CI 2-sided [0.83 to 1.64]

ADVERSE EVENTS:
Description: 128 participants in Placebo as 1 participant withdrew consent prior to treatment
Arm/Group | Olaparib 400 mg bd | Placebo
Serious Adverse Events (participants affected / at risk) | 31/136 | 11/128
Other Adverse Events (participants affected / at risk) | 129/136 | 111/128
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Olaparib 400 mg bd (N=136) | Placebo (N=128)
ANAEMIA (Blood and lymphatic system disorders) | 3 (3) | 0 (0)
PANCYTOPENIA (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
CARDIOVASCULAR INSUFFICIENCY (Cardiac disorders) | 1 (1) | 0 (0)
ABDOMINAL INCARCERATED HERNIA (Gastrointestinal disorders) | 1 (1) | 0 (0)
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 (0) | 1 (2)
CONSTIPATION (Gastrointestinal disorders) | 2 (2) | 0 (0)
DIARRHOEA (Gastrointestinal disorders) | 1 (1) | 0 (0)
GASTRITIS (Gastrointestinal disorders) | 0 (0) | 2 (2)
IMPAIRED GASTRIC EMPTYING (Gastrointestinal disorders) | 0 (0) | 1 (1)
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1 (1) | 1 (1)
INTRA-ABDOMINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 0 (0)
MELAENA (Gastrointestinal disorders) | 1 (1) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 1 (1) | 0 (0)
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 2 (2) | 3 (4)
VOMITING (Gastrointestinal disorders) | 1 (1) | 0 (0)
HERNIA PAIN (General disorders) | 1 (1) | 0 (0)
NON-CARDIAC CHEST PAIN (General disorders) | 1 (1) | 0 (0)
PYREXIA (General disorders) | 1 (1) | 0 (0)
IODINE ALLERGY (Immune system disorders) | 1 (1) | 0 (0)
APPENDICITIS (Infections and infestations) | 1 (1) | 0 (0)
ENDOPHTHALMITIS (Infections and infestations) | 0 (0) | 1 (1)
INFECTIVE EXACERBATION OF CHRONIC OBSTRUCTIVE AIRWAYS DISEASE (Infections and infestations) | 0 (0) | 1 (1)
INFLUENZA (Infections and infestations) | 0 (0) | 1 (1)
LIVER ABSCESS (Infections and infestations) | 1 (1) | 0 (0)
PNEUMONIA (Infections and infestations) | 1 (1) | 0 (0)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 (1) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 1 (1) | 1 (1)
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
HIP FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
POST PROCEDURAL HAEMATOMA (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
DEHYDRATION (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
OSTEOPOROSIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
ACUTE LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
BLADDER CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
INTRADUCTAL PROLIFERATIVE BREAST LESION (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
PAPILLARY THYROID CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
SQUAMOUS CELL CARCINOMA OF THE ORAL CAVITY (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
APHASIA (Nervous system disorders) | 1 (1) | 0 (0)
HAEMORRHAGIC STROKE (Nervous system disorders) | 1 (1) | 0 (0)
SYNCOPE (Nervous system disorders) | 1 (1) | 0 (0)
CONFUSIONAL STATE (Psychiatric disorders) | 1 (1) | 0 (0)
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
BRONCHIECTASIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
COUGH (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
DEEP VEIN THROMBOSIS (Vascular disorders) | 1 (1) | 0 (0)
ESSENTIAL HYPERTENSION (Vascular disorders) | 0 (0) | 1 (1)
VENA CAVA THROMBOSIS (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Olaparib 400 mg bd (N=136) | Placebo (N=128)
ANAEMIA (Blood and lymphatic system disorders) | 26 (32) | 7 (8)
NEUTROPENIA (Blood and lymphatic system disorders) | 7 (8) | 5 (7)
ABDOMINAL DISCOMFORT (Gastrointestinal disorders) | 6 (7) | 7 (7)
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 21 (24) | 11 (13)
ABDOMINAL PAIN (Gastrointestinal disorders) | 35 (44) | 34 (51)
ABDOMINAL PAIN LOWER (Gastrointestinal disorders) | 7 (7) | 10 (10)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 25 (28) | 11 (11)
CONSTIPATION (Gastrointestinal disorders) | 30 (41) | 14 (15)
DIARRHOEA (Gastrointestinal disorders) | 36 (62) | 31 (39)
DYSPEPSIA (Gastrointestinal disorders) | 27 (34) | 11 (11)
NAUSEA (Gastrointestinal disorders) | 96 (128) | 46 (58)
STOMATITIS (Gastrointestinal disorders) | 12 (15) | 4 (4)
VOMITING (Gastrointestinal disorders) | 47 (91) | 18 (20)
ASTHENIA (General disorders) | 19 (26) | 12 (15)
FATIGUE (General disorders) | 73 (92) | 50 (57)
OEDEMA PERIPHERAL (General disorders) | 12 (14) | 6 (7)
PYREXIA (General disorders) | 13 (16) | 4 (4)
NASOPHARYNGITIS (Infections and infestations) | 21 (26) | 14 (17)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 18 (24) | 8 (8)
URINARY TRACT INFECTION (Infections and infestations) | 15 (21) | 6 (6)
BLOOD CREATININE INCREASED (Investigations) | 9 (10) | 2 (2)
DECREASED APPETITE (Metabolism and nutrition disorders) | 29 (34) | 17 (22)
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 8 (10) | 9 (10)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 24 (36) | 18 (19)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 25 (37) | 14 (16)
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 13 (20) | 5 (5)
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 10 (10) | 8 (8)
MYALGIA (Musculoskeletal and connective tissue disorders) | 7 (7) | 8 (9)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 12 (16) | 7 (8)
DIZZINESS (Nervous system disorders) | 21 (28) | 9 (10)
DYSGEUSIA (Nervous system disorders) | 22 (26) | 8 (8)
HEADACHE (Nervous system disorders) | 29 (47) | 17 (20)
NEUROPATHY PERIPHERAL (Nervous system disorders) | 12 (13) | 3 (5)
PARAESTHESIA (Nervous system disorders) | 7 (9) | 3 (5)
ANXIETY (Psychiatric disorders) | 8 (8) | 5 (6)
DEPRESSION (Psychiatric disorders) | 11 (11) | 9 (10)
INSOMNIA (Psychiatric disorders) | 9 (9) | 9 (10)
COUGH (Respiratory, thoracic and mediastinal disorders) | 23 (33) | 13 (14)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 17 (20) | 8 (8)
DRY SKIN (Skin and subcutaneous tissue disorders) | 3 (3) | 7 (7)
PRURITUS (Skin and subcutaneous tissue disorders) | 8 (10) | 3 (3)
RASH (Skin and subcutaneous tissue disorders) | 8 (8) | 12 (13)
HOT FLUSH (Vascular disorders) | 5 (6) | 16 (18)
HYPERTENSION (Vascular disorders) | 10 (10) | 4 (4)

LIMITATIONS AND CAVEATS:
For OM DoR: The subset of patients evaluable for response who responded to study treatment.Values in results table may be under-estimates as some patients had not progressed at final analysis,so true duration is likely to be greater than in database.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less